CLINICAL TRIAL: NCT03870555
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, 3-Period, Incomplete Block Design Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-954 in Healthy Adult Participants
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of TAK-954 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: TAK-954-1009; U1111-1224-9803 (Registry Identifier: WHO)
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): Period 1: TAK-954 placebo-matching infusion, administered intravenously over 60-minutes, once on Day 1 and Day 2.
  Period 2: TAK-954 0.1 milligram (mg), infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 1 mg infusion, administered intravenously over 60-minutes, once on Day 2.
  Period 3: TAK-954 0.1 mg, infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 2 mg infusion, administered intravenously over 60-minutes, once on Day 2.
  A washout period of at least 16 days will be maintained between each Treatment Period.
  Interventions: Drug: TAK-954; Drug: TAK-954 Placebo
- Sequence 2 (Experimental): Period 1: TAK-954 0.1 mg, infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 0.5 mg infusion, administered intravenously over 60-minutes once on Day 2.
  Period 2: TAK-954 placebo-matching infusion, administered intravenously over 60-minutes, once on Day 1 and Day 2.
  Period 3: TAK-954 0.1 mg, infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 2 mg, infusion, administered intravenously over 60-minutes, once on Day 2.
  A washout period of at least 16 days will be maintained between each Treatment Period.
  Interventions: Drug: TAK-954; Drug: TAK-954 Placebo
- Sequence 3 (Experimental): Period 1: TAK-954 0.1 mg, infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 0.5 mg, infusion, administered intravenously over 60-minutes once on Day 2.
  Period 2: TAK-954 0.1 mg, infusion, administered intravenously over 60-minutes, once on Day 1, TAK-954 1 mg, infusion, administered intravenously over 60-minutes, once on Day 2.
  Period 3: TAK-954 placebo-matching infusion, administered intravenously over 60-minutes, once on Day 1 and Day 2. A washout period of at least 16 days will be maintained between each Treatment Period.
  Interventions: Drug: TAK-954; Drug: TAK-954 Placebo

INTERVENTIONS:
Drug: TAK-954 — TAK-954 infusion administered intravenously.
Drug: TAK-954 Placebo — TAK-954 placebo-matching infusion intravenous.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of single ascending intravenous doses of TAK-954.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. This study will assess the safety, tolerability, PK and PD of single ascending TAK-954 higher intravenous doses than those previously studied.

The study will enroll approximately 6 participants. Participants will be randomly assigned (By chance, like flipping a coin) to one of the three treatment sequences-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

In each treatment sequence, each participant will receive 2 doses of active drug out of 3 dose levels (TAK-954 0.5 mg, TAK-954 1 mg, or TAK-954 2 mg) and 1 dose of Placebo. Dose escalation will be based on the available safety/tolerability data from the previous period.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 73 days. Participants will make a final visit on Day 16 after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 32 kilogram per square meter (kg/m^2), weighing >=50 kilogram (kg) at screening.
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, orthostatic vital signs, or ECGs, as deemed by the Investigator or designee.
3. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study, based on participant self-reporting.

Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
2. Has infrequent bowel movements (less than approximately once per day) within 30 days prior to first dosing.
3. Recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 2 weeks of first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 08 March 2019 to 16 May 2019.
Pre-assignment Details: Healthy adult participants were enrolled in this 3-period cross-over study in 1 of the 3 treatment sequences to receive TAK-954 0.1 milligram (mg) or Placebo on Day 1 (Lead-in Dose), followed by TAK-954 (0.5 mg, 1 mg or 2 mg) or Placebo on Day 2 (Treatment Dose) of each study period.
Groups:
- Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg: Period 1: TAK-954 placebo-matching infusion, intravenously, once on Day 1 and Day 2.
  Period 2: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 1 mg infusion, intravenously, once on Day 2.
  Period 3: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 2 mg infusion, intravenously, once on Day 2.
  A washout period of at least 16 days was maintained between each Treatment Period.
- Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg: Period 1: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 0.5 mg infusion, intravenously once on Day 2.
  Period 2: TAK-954 placebo-matching infusion, intravenously, once on Day 1 and Day 2.
  Period 3: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 2 mg, infusion, intravenously, once on Day 2.
  A washout period of at least 16 days was maintained between each Treatment Period.
- Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo: Period 1: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 0.5 mg, infusion, intravenously once on Day 2.
  Period 2: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 and TAK-954 1 mg, infusion, intravenously, once on Day 2.
  Period 3: TAK-954 placebo-matching infusion, intravenously, once on Day 1 and Day 2.
  A washout period of at least 16 days was maintained between each Treatment Period.
Period: Period 1 (2 Days)
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Washout Period (at Least 16 Days)
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Washout Period (at Least 16 Days)
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Period 3 (2 Days)
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo
Started | 2 | 2 | 2
Completed | 1 | 2 | 2
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of the study drug (active or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Placebo + TAK-954 1 mg + TAK-954 2 mg | Sequence 2: TAK-954 0.5 mg + Placebo + TAK-954 2 mg | Sequence 3: TAK-954 0.5 mg + TAK-954 1 mg + Placebo | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (14.14) | 33.0 (4.24) | 46.5 (2.12) | 35.8 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 2 | 6
Weight [Mean (Standard Deviation); unit: kilogram] | 84.80 (13.152) | 67.60 (9.758) | 80.55 (0.495) | 77.65 (10.858)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.5 (7.78) | 167.0 (21.21) | 165.5 (4.95) | 167.0 (10.43)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.655 (1.9021) | 24.375 (2.5102) | 29.455 (1.7607) | 27.828 (3.1252)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) for TAK-954
Time Frame: Dosing on Day 2 in Period 1 up to 14 days after last dose of study drug on Day 2 of Period 3 (up to Day 52)
Population: The safety set included all participants who received at least one dose of the study drug (active or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Dose: TAK-954 0.5 mg: TAK-954 0.5 mg, infusion, intravenously, once on Day 2 of Period 1 in Sequence 2 or 3.
- Treatment Dose: TAK-954 1 mg: TAK-954 1 mg, infusion, intravenously, once on Day 2 of Period 2 in Sequence 1 or 3.
- Treatment Dose: TAK-954 2 mg: TAK-954 2 mg, infusion, intravenously, once on Day 2 of Period 3 in Sequence 1 or 2.
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 4 | 3 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs for TAK-954
Time Frame: Dosing on Day 2 in Period 1 up to 14 days after last dose of study drug on Day 2 of Period 3 (up to Day 52)
Population: The safety set included all participants who received at least one dose of the study drug (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiograms (ECG) for TAK-954
Time Frame: Dosing on Day 2 in Period 1 up to 14 days after last dose of study drug on Day 2 of Period 3 (up to Day 52)
Population: The safety set included all participants who received at least one dose of the study drug (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Notable Shifts From Baseline to Abnormal Post-dose in Clinical Laboratory Values for TAK-954
Time Frame: Dosing on Day 2 in Period 1 up to 14 days after last dose of study drug on Day 2 of Period 3 (up to Day 52)
Population: The safety set included all participants who received at least one dose of the study drug (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 0 | 0 | 0

5. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*hr/mL)
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
picogram*hour per milliliter (pg*hr/mL) | 88930 (23.0) | 163200 (12.8) | 298400 (29.6)

6. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
pg*hr/mL | 89220 (22.8) | 163700 (12.8) | 299500 (29.6)

7. Primary Outcome: Ceoi: Plasma Concentration Observed at the End of Infusion for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
picogram per milliliter (pg/mL) | 7502 (24.1) | 15260 (12.9) | 30270 (28.5)

8. Primary Outcome: CL: Total Clearance After Intravenous Administration for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
liter per hour (L/hr) | 5.604 (22.8) | 6.110 (12.8) | 6.679 (29.6)

9. Primary Outcome: Vz: Volume of Distribution During the Terminal Disposition Phase After Intravenous Administration for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
liter | 197.9 (13.7) | 387.7 (45.6) | 901.7 (61.7)

10. Primary Outcome: Ae: Amount of Unchanged Drug Excreted in the Urine for TAK-954 on Day 2 up to 12 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
nanogram | 104300 (6.3) | 226000 (16.0) | 408900 (15.3)

11. Primary Outcome: Ae: Amount of Unchanged Drug Excreted in the Urine for TAK-954 on Day 2 up to 24 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations). PK-evaluable population where data at specified time points was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
nanogram | 53200 (27.3) | 115300 (19.9) | 190700 (23.7)

12. Primary Outcome: Ae: Amount of Unchanged Drug Excreted in the Urine for TAK-954 on Day 2 up to 36 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
nanogram | 32420 (17.3) | 66560 (5.3) | 103600 (8.5)

13. Primary Outcome: Fe: Fraction of TAK-954 Excreted in Urine on Day 2 up to 12 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
percentage | 20.86 (6.3) | 22.60 (16.0) | 20.45 (15.3)

14. Primary Outcome: Fe: Fraction of TAK-954 Excreted in Urine on Day 2 up to 24 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
percentage | 10.64 (27.3) | 11.53 (19.9) | 9.534 (23.7)

15. Primary Outcome: Fe: Fraction of TAK-954 Excreted in Urine on Day 2 up to 36 Hours Post-dose
Time Frame: Day 2 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
percentage | 6.484 (17.3) | 6.656 (5.3) | 5.181 (8.5)

16. Primary Outcome: CLR: Renal Clearance for TAK-954
Time Frame: Day 2 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 3 | 4 | 3
L/hr | 3.457 (19.9) | 3.933 (8.9) | 3.624 (35.0)

17. Secondary Outcome: Number of Participants With First Stool of TAK-954 Within 36 Hours Post-dose on Day 2
Time Frame: Day 2 dosing and at multiple time points (up to 36 hours) post-dose
Population: The pharmacodynamic (PD) set included all participants who received at least one dose of the study drug (active or placebo) and had completed at least 1 PD sampling period and/or had at least 1 evaluable parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 3 | 4 | 3

18. Secondary Outcome: Mean Number of Stools of TAK-954 Within 36 Hours Post-dose on Day 2
Time Frame: Day 2 dosing and at multiple time points (up to 36 hours) post-dose
Population: The PD set included all participants who received at least one dose of the study drug (active or placebo) and had completed at least 1 PD sampling period and/or had at least 1 evaluable parameter.
Measure: Mean (Standard Deviation); unit: stools
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
stools | 3.3 (3.40) | 2.0 (0.82) | 1.0 (0.00)

19. Secondary Outcome: Instances of Stool Type of TAK-954 Based on Bristol Stool Form Scale
Description: Number of occurrences for each stool type was reported based on their type assessed from Bristol Stool form scale. The Bristol Stool Form Scale was used to assess the stool shape using a 7-point scale. Where, Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid. A score of 1 or 2 indicates constipation and a score of 6 or 7 indicates diarrhea.
Time Frame: Day 2 dosing and at multiple time points (up to 36 hours) post-dose
Population: as for outcome 18
Measure: Number; unit: number of occurrences
Arm/Group | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg
Number analyzed (Participants) | 4 | 4 | 3
number of occurrences
  Type 1 | 0 | 0 | 0
  Type 2 | 2 | 3 | 2
  Type 3 | 0 | 1 | 0
  Type 4 | 1 | 2 | 1
  Type 5 | 3 | 1 | 0
  Type 6 | 5 | 1 | 0
  Type 7 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Lead-in Dose: Day 1 of Period 1, 2, and 3; Treatment Dose: Dosing on Day 2 in Period 1 up to 14 days after last dose of study drug on Day 2 of Period 3 (up to Day 52)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Lead-in Dose: TAK-954 0.1 mg: TAK-954 0.1 mg, infusion, intravenously, once on Day 1 of Period 1, 2 or 3 in Sequence 1, 2, or 3.
- Lead-in Dose: Placebo: TAK-954 placebo-matching, infusion, intravenously, once on Day 1 of Period 1, 2, or 3 in Sequence 1, 2, or 3.
- Treatment Dose: Placebo: TAK-954 placebo-matching, infusion, intravenously once on Day 2 of Period 1, 2 and 3.
Arm/Group | Lead-in Dose: TAK-954 0.1 mg | Lead-in Dose: Placebo | Treatment Dose: TAK-954 0.5 mg | Treatment Dose: TAK-954 1 mg | Treatment Dose: TAK-954 2 mg | Treatment Dose: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 1/6 | 4/4 | 3/4 | 0/3 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Dose: TAK-954 0.1 mg (N=6) | Lead-in Dose: Placebo (N=6) | Treatment Dose: TAK-954 0.5 mg (N=4) | Treatment Dose: TAK-954 1 mg (N=4) | Treatment Dose: TAK-954 2 mg (N=3) | Treatment Dose: Placebo (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03870555/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03870555/SAP_001.pdf